CLINICAL TRIAL: NCT03067207
Title: A Randomized-Control Trial of an In-Person vs e-Health Mindfulness-Based Intervention for Adolescents With Chronic Illness
Brief Title: In-Person vs e-Health Mindfulness-Based Intervention for Adolescents With Chronic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Mind and Life Institute, Hadley, Massachusetts (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Miriam Kaufman, Division Head, Adolescent Medicine, The Hospital for Sick Children
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: REB1000053600
Record Dates: First submitted 2017-02-15; First posted 2017-03-01 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Chronic Illness; Mental Health Impairment
Keywords: mindfulness meditation; Adolescent; eHealth; randomized trial
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a longitudinal randomized non-inferiority trial comparing two arms: an experimental arm and feasibility arm. Participants living close enough to commit to in-person sessions will be entered in the experimental arm of the study. The feasibility arm, which will only take place if the targeted number of study participants (60) is not reached for the experimental arm, will be offered to participants who are not able to commit to the in-person mode of delivery. It will consist of two groups, one early e-health group and one wait-list e-Health group. At the end of the recruitment period, once participants have been placed in the experimental and feasibility arms, two separate randomizations will take place. The first randomization (experimental arm) will serve to assign participants to one of the four experimental groups and the second randomization (feasibility arm) will assign participants to one of the two feasibility groups.
Who Masked: Investigator
Masking Description: This study will be a single-blinded study (investigators only). Participants will be coded using Arabic numerals. A research assistant will receive all questionnaires and cortisol samples. Mindfulness facilitators will be unaware of participant identification numbers. Participants will be assigned to one of four groups (experimental arm) or to one of two groups (feasibility arm) following a computer-generated randomization list (permuted block design, using blocks of two or four). The allocation sequence will be generated by a statistician not otherwise involved in the project and passed on to a research assistant after patient identification data has been collected (ensuring that the investigators are kept blind to the allocation of each participant). Allocation sequence will be password-protected and only accessible by the statistician and research assistant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental arm will consist of four groups with a target of 15 participants each: one early intervention group, one wait-list in-person group, one early e-Health group and one wait-list e-health group. All participants will receive the mindfulness intervention, MARS-A, either in-person or via e-health by the end of the 6-month study period. Participants in the in-person groups will meet at in hospital at a designated teen-friendly room containing chairs and yoga mats. Participants in the e-health groups will be encouraged to find a quiet room in their home and will be required to have access to the Internet, a desktop/laptop computer equipped with a webcam or a tablet/smartphone with webcam function.
  Interventions: Behavioral: MARS-A
- Feasibility (Other): The feasibility arm, which will only take place if the targeted number of study participants (60) is not reached for the experimental arm, will be offered to participants who are not able to commit to the in-person mode of delivery. It will consist of two groups, one early e-health group and one wait-list e-Health group. The intervention delivered, MARS-A, will be identical as the intervention delivered to e-health groups in the experimental arm.
  Interventions: Behavioral: MARS-A

INTERVENTIONS:
Behavioral: MARS-A — The intervention will consist of the 8-week mindfulness meditation program designed for adolescents with chronic health conditions.MARS-A is based on two established mindfulness-based interventions for adults: MBSR and MBCT. The content of the program will be the same for in-person and e-health groups: all participants will receive eight 90-minute weekly evening sessions led by two trained and experienced mindfulness providers. Sessions will include short meditation practices, breathing exercises, guided discussion, mindful movements and inquiry, adapted to the context of chronic illness. Every session will start with a brief review of home practice and will close with a discussion of the home practice for the following week.
  Other Names: Mindful Awareness and Resiliency Skills for Adolescents

SUMMARY:
This study will seek to compare the effect of a mindfulness meditation program for adolescents with chronic illness delivered either in person or via an online platform. The 8-week program will combine meditation practices, breathing exercises and group discussions. Participants will be recruited from different general and specialized clinics at the Hospital for Sick Children and will be allocated to either an in-person or the online group through a random process (like tossing a coin). The study will aim to recruit 60 participants ages 13-18. Each participant will provide data through research questionnaires, recorded interviews and saliva samples.

DETAILED DESCRIPTION:
The study will be conducted as a longitudinal randomized controlled trial comparing in-person and eHealth delivery of a mindfulness meditation intervention for adolescents with chronic illness. There will be two arms. An experimental and a feasibility arm. In the experimental arm, 4 groups of 10-15 participants will be formed: two in-person groups (early and late) and two eHealth groups (early and late). The early groups will receive the intervention at the beginning of the study period and the late groups will be wait-list controlled group that will receive the intervention at the middle of the study period. At the end of the recruitment period or when the target number of participants is met (60), whichever comes first, all teens meeting the inclusion criteria will be randomly allocated to one of the four randomized groups. Teens who are not meeting the final inclusion criteria (able to attend mindfulness sessions at Sickkids) will be offered a spot in the feasibility arm of the study until the maximum total number of study participants is reached (60). These participants will be placed in eHealth groups (either early or late) through a separate randomization process.

Data collection will take place at baseline (during the intake meeting), immediately before and following the mindfulness intervention as well as at the end of the 6-month study period. Participants in the experimental arm will provide data through research questionnaires, salivary cortisol analysis as well as individual semi-structured interviews with a research assistant. Salivary samples will be provided from home for participants in the eHealth groups. Participants in the feasibility arm will only provide information through research questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic illness
* Fluent in English
* Followed by a care provider at the Hospital for SickKids
* Able to consent to the study
* Able to attend in-person mindfulness meditation sessions at Sickkids (for the experimental arm only)

Exclusion Criteria:

* Active and unaddressed suicidal ideation
* Developmental disability preventing participation in the mindfulness program

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Mindfulness Skills Acquisition | Up to 6 months
  Acquisition of mindfulness skills as measured by the MAAS-A questionnaire a 14-item Likert-type scale that has been validated in adolescents.

SECONDARY OUTCOMES:
Anxiety and depression score | Up to 6 months
  Anxiety and depression scores as measured by the DASS-21 questionnaire, a Likert-type scale that has been validated in adolescents
Self-Esteem | Up to 6 months
  Self-esteem scores as measured by the Rosemberg Self-Esteem Scale a validated Likert-type scale that has been validated in adolescents.
Salivary cortisol levels | Up to 6 months
  Salivary cortisol levels measured at 8am, 12pm, pre and post meditation at weeks 1 and 8 of the intervention. Sampled by Salivette devices (cotton swabs) and analyzed by enzyme immune-assay
Perception of Illness | Up to 6 months
  Perception of illness score (coping with chronic health condition) as measured by the Perceptions of Illness questionnaires a validated Likert-type scale.
Mindfulness home-practice | Up to 6 months
  Compilation of personal mindfulness meditation practice through self-reported log books filled at the beginning of each session of the 8-week mindfulness meditation program.
Appreciation of the mindfulness intervention | Up to 6 months
  Semi-structured interviews conducted by research assistant with participants having completed the 8-week mindfulness meditation program. Interviews will compare appreciation between in-person and e-Health groups

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kaufman, MD, Principal Investigator — Hospital for Sickkids

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chadi N, McMahon A, Vadnais M, Malboeuf-Hurtubise C, Djemli A, Dobkin PL, Lacroix J, Luu TM, Haley N. Mindfulness-based Intervention for Female Adolescents with Chronic Pain: A Pilot Randomized Trial. J Can Acad Child Adolesc Psychiatry. 2016 Fall;25(3):159-168. Epub 2016 Nov 1. PMID 27924146
- [Derived] Chadi N, Kaufman M, Weisbaum E, Malboeuf-Hurtubise C, Kohut SA, Viner C, Locke J, Vo DX. In-Person Versus eHealth Mindfulness-Based Intervention for Adolescents With Chronic Illness: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Nov 27;6(11):e241. doi: 10.2196/resprot.7700. PMID 29180345